CLINICAL TRIAL: NCT02570672
Title: Metformin for Preventing Frailty in High-risk Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sara E Espinoza, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSC20150237H; 1R01AG052697-01A1 (NIH)
Record Dates: First submitted 2015-09-08; First posted 2015-10-07 (Estimated); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-05

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Subjects will be randomized to metformin (titrated up to 1000 mg twice daily, as tolerated)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Subjects will be randomized to metformin (titrated up to 1000 mg twice daily, as tolerated) vs. placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Subjects will be randomized to metformin titrated to 1000mg twice daily as tolerated.
  Arms: Metformin
Drug: Placebo — Subjects will randomized to placebo will receive placebo
  Arms: Placebo

SUMMARY:
Frailty is a geriatric syndrome which leads to poor health outcomes in older adults, such as falls, disability, hospitalization, institutionalization, and death. Due to the dramatic growth in the U.S. aging population and the health care costs associated with frailty (estimated at more than $18 billion per year), frailty is a major health care problem. There has been little research into potential pharmacologic interventions that would delay or reduce the incidence of frailty. Thus, the major goal of this study is to test metformin as a novel intervention for the prevention of frailty. The investigators propose that diabetes/insulin resistance and inflammation are major contributors to frailty, and that the use of metformin to modulate diabetes/insulin resistance and inflammation will prevent and/or ameliorate the progression of frailty.

DETAILED DESCRIPTION:
Physical frailty is a geriatric syndrome that leads to poor health outcomes such as falls, disability, institutionalization, and death. The prevalence of frailty is estimated to be 7-15% among community-dwelling older U.S. adults. The associated costs of frailty were estimated to be more than $18 billion in 2000 and these will continue to increase over the next two decades. Thus, an increasingly frail older population will have major implications for the demand for health care services, including hospital usage, home care, and long-term care.

Data from several studies have suggested strong roles for diabetes and insulin resistance, which are associated with increased inflammation, in the physiological basis of frailty. The investigators' recent epidemiological research with a community-based population of older adults showed that diabetes was the most significant predictor of frailty onset and worsening over time. While the importance of frailty and its impact on an aging U.S. society have been widely recognized, to date there are no effective interventions to prevent or treat frailty. Therefore, the major goal of this study is to test a drug with insulin-sensitizing and anti-inflammatory properties, such as metformin, as a novel intervention for frailty prevention.

The investigators hypothesize that metformin will lead to reduced inflammation and insulin resistance present in older glucose-intolerant subjects and that these changes will consequently prevent the onset and/or progression of frailty in this sub-population of older adults. Subjects with impaired glucose intolerance will be enrolled in this study because this group encompasses approximately 1/3rd of the older population, this group is at increased risk for developing diabetes and frailty, and is the most likely to benefit from a potential anti-inflammatory and insulin-sensitizing intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* All ethnic groups
* Age 65 and older
* Community-dwelling
* Pre-diabetic based on oral glucose tolerance test with 2 hour values of 140 - 199 mg/dL after an oral glucose load, and no diagnosis of diabetes in the past 12 months
* Subjects must have the following laboratory values: Hematocrit ≥ 33%, aspartate aminotransferase < 2 X upper limit of normal, alanine aminotransferase < 2 X upper limit of normal, alkaline phosphatase < 2 X upper limit of normal, normal urinalysis (no clinically significant white blood cells, red blood cells or bacteria), platelets ≥ 100,000, prothrombin time < 15 seconds and partial thromboplastin time < 40 seconds, glomerular filtration rate (GFR) ≥ 45ml/min and urine protein ≤ 100 mg/dL by lab urinalysis.

Exclusion Criteria:

* Characterized as frail, defined as the presence of 3 or more of: 1) weak hand grip strength, 2) slow walking speed, 3) low physical activity, 4) unintentional weight loss of ≥ 10 pounds over the past year, 5) self-reported exhaustion
* Resident of nursing home or long-term care facility
* Subjects with diabetes with range fasting glucose in diabetes range (≥ 126 mg/dL), or 2-hour glucose within diabetes range on OGTT (≥ 200 mg/dL).
* Subjects taking drugs known to affect glucose homeostasis
* Untreated depression or Geriatric Depression Scale (GDS) score on 15-item scale >7
* Diagnosis of any disabling neurologic disease Parkinson's Disease, Amyotrophic Lateral Sclerosis, multiple sclerosis, cerebrovascular accident with residual deficits (muscle weakness or gait disorder), severe neuropathy, diagnosis of dementia or Mini-mental State Exam (MMSE) score <24, cognitive impairment due to any reason such that the patient is unable to provide informed consent.
* History of moderate-severe heart disease (New York Heart Classification greater than grade II) or pulmonary disease (dyspnea on exertion upon climbing one flight of stairs or less; abnormal breath sounds on auscultation)
* Poorly controlled hypertension (systolic >160 mmHg, diastolic >100 mmHg)
* Peripheral arterial disease (history of claudication)
* Moderate to severe valvular heart disease
* Subjects who have been treated with long term (>30 days) systemic steroids, anabolic steroids, growth hormone or immunosuppresants within the last 6 months. Males with a medical history of testosterone deficiency who are on a stable dose of testosterone replacement (for ≥ 3 months) are allowed.
* Subjects who have been treated with short term (<30 days) systemic steroids, anabolic steroids, growth hormone or immunosuppressants within the last 1 month.
* Chronic inflammatory condition, autoimmune disease, or infectious processes (e.g., active tuberculosis, Human Immunodeficiency Virus, rheumatoid arthritis, systemic lupus erythematosus, acute or chronic hepatitis B or C)
* Active tobacco use (within 6 months)
* Illicit drug use
* Active malignancy, non-skin
* Disease or condition likely to cause death within 5 years
* Hypersensitivity to metformin or pioglitazone
* Any disease or condition considered to be exclusionary based on the clinical opinion and discretion of the PI

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara E Espinoza, M.D., Principal Investigator — Associate Professor
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 70 | 71
Completed | 58 | 67
Not Completed | 12 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 70 | 71 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (5.4) | 72.6 (5.1) | 71.78 (5.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 36 | 37 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 22 | 49
  Not Hispanic or Latino | 43 | 49 | 92
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 64 | 68 | 132
  African American | 3 | 3 | 6
  Other | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 70 | 71 | 141

OUTCOME MEASURES:

1. Primary Outcome: Frailty Index Based on Deficit Accumulation
Description: Frailty index based on deficit accumulation. The frailty index will be measured based on the presence of several potential deficits, including chronic diseases, conditions, and impairments. Deficits are ascertained from study visit assessments, including medical history, physical examination, physical function, cognitive function, disability, and quality of life. The frailty index score was calculated as the ratio of the number of deficits to the total number of deficits. The total range of the index is 0 to 1, with higher score indicating more frailty. The outcome is the covariate adjusted monthly rate of change in the frailty index over the study period.
Time Frame: 2 years
Population: Participants that completed study
Measure: Mean (Standard Error); unit: Index score
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 58 | 67
Index score | -0.0002 (0.0002) | 0.0002 (0.0002)

2. Primary Outcome: Fried Frailty Phenotype Criteria
Description: The frailty score will be measured based on the following 5 frailty characteristics: 1) unintentional weight loss of >= 10 pounds in last year at baseline and ≥5% loss of body weight during follow-up; 2) self-reported exhaustion based on the Geriatric Depression Scale item, "Do you feel full of energy?;" 3) muscle weakness based on hand grip strength measurement (standardized cut points are published); 4) slow gait speed based on 10-foot walk (standardized cut points are published); and 5) low physical activity measured in kilocalories/week based on the Minnesota Leisure Time Questionnaire (standardized cut points are published). The Fried frailty score was calculated as the number of frailty characteristics present, each with a score of 0 or 1. The total range of scores is 0-5, with a higher score indicating more frailty. The outcome is the covariate adjusted monthly rate of change in the Fried frailty score over the study period.
Time Frame: Baseline to 2 years
Population: Participants that completed the study
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 58 | 67
Score on a scale | 0.0289 (0.0049) | 0.0164 (0.0058)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to 2 years.
Description: All cause mortality and serious adverse events, related and unrelated to study intervention, are reported.
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 1/71
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/71
Other Adverse Events (participants affected / at risk) | 70/70 | 71/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=70) | Placebo (N=71)
Diarrhea (Gastrointestinal disorders) | 50 (133) | 33 (75)
Arthralgia (Nervous system disorders) | 22 (33) | 24 (55)
Nausea (Gastrointestinal disorders) | 21 (31) | 12 (18)
Flatulence (Gastrointestinal disorders) | 15 (22) | 7 (11)
Peripheral edema (Blood and lymphatic system disorders) | 15 (21) | 13 (16)
Pain in extremity (General disorders) | 15 (19) | 15 (26)
Contusion (Blood and lymphatic system disorders) | 14 (21) | 17 (26)
Headache (Nervous system disorders) | 14 (23) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/72/NCT02570672/Prot_SAP_000.pdf